CLINICAL TRIAL: NCT05477121
Title: Severity: Quantifying the Severity of Generalized Tonic-clonic Seizures (GTCS) With Connected Devices
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Philippe Ryvlin, Professor, head of the department of clinical neurosciences, principal investigator, Centre Hospitalier Universitaire Vaudois
Other Study IDs: SEVERITY
Record Dates: First submitted 2022-03-12; First posted 2022-07-28 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Epilepsy, Generalized
MeSH Terms: conditions — Epilepsy, Generalized

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
By bringing together the fields of seizure detection and that of Sudden Unexpected Death in Epilepsy (SUDEP), the current project aims at delineating which set of biosensors and related biomarkers would optimally characterize the severity of GTCS and the associated risk of SUDEP.

DETAILED DESCRIPTION:
The main objective is to to evaluate which of the five biosignals considered, being, electrodermal activity (EDA), heart rate (HR), accelerometry (AC), arm-measurement of skin electromyography (EMG), and bed sensing of body movement (BM), or any of their combinations, offers the most accurate detection and quantification of our primary indicator of GTCS-severity, i.e. postictal EEG suppression (PGES).

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 12 years or older, suffering from epilepsy
* Patient undergoing Video-EEG recording
* Patient at risk of presenting a GTCS during Video-EEG monitoring according to one of the following criteria (i) known to suffer from GTCS, or (ii) considered for Antiepileptic drugs (AED) tapering during Video-EEG (GTCS often occur during Video-EEG as a result of AED tapering for promoting the occurrence of seizures).
* Patient willing to participate in the study and signed informed consent, by patient or legal representative when required.

Exclusion Criteria:

* Patients aged less than 12 years old
* Patient not willing to participate in the study, and where informed consent from the patient or the legal representative, when required, cannot be obtained - Patient considered not at risk of presenting a GTCS during Video-EEG because they are not known to suffer GTCS and not candidate to AED tapering during Video-EEG.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A cohort of 500 patients with active epilepsy, undergoing Video-EEG monitoring in one of the participating epilepsy centers will be enrolled in this study with the aim to record epileptic seizures for routine clinical, and not primarily research objectives (e.g. presurgical evaluation, other diagnostic purposes). The project population will be composed of adult patients who give informed consent independently as well as of children, and adult patients who lack the capacity to consent to matters concerning their personal health care.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
duration of PGES | Through study completion, an average of 4 years
  The primary endpoint of the study is the duration of PGES, as defined by a postictal EEG flattening <10microvolt over all scalp-EEG leads (time in seconds). When no PGES is observed, the duration will be coded as 0. This will be used as a dependent variable in the primary analysis.

SECONDARY OUTCOMES:
Type of GTCS | Through study completion, an average of 4 years
  According to our previously published classification.
GTCS tonic phase duration on video-EEG recording | Through study completion, an average of 4 years
  In seconds
GTCS clonic phase duration on video-EEG recording | Through study completion, an average of 4 years
  In seconds
Postictal upper limb immobility duration on video-EEG recording | Through study completion, an average of 4 years
  In seconds
Postictal whole-body immobility duration on video-EEG recording | Through study completion, an average of 4 years
  In seconds
Postictal confusion duration on video-EEG recording | Through study completion, an average of 4 years
  In seconds
Postictal bradycardia presence on Electrocardiogram (EKG) | Through study completion, an average of 4 years
  Yes or No
Postictal bradycardia duration on EKG | Through study completion, an average of 4 years
  In seconds
Postictal bradycardia nadir on EKG | Through study completion, an average of 4 years
  Heart rate per minute
Postictal hypoxemia presence on pulse oxymetry | Through study completion, an average of 4 years
  Yes or No
Postictal hypoxemia duration on pulse oxymetry | Through study completion, an average of 4 years
  In seconds
Postictal hypoxemia nadir | Through study completion, an average of 4 years
  Spo2 value in %
Peri-ictal tachycardia or bradycardia presence | Through study completion, an average of 4 years
  Yes or No
Peri-ictal tachycardia or bradycardia duration | Through study completion, an average of 4 years
  In seconds
Peri-ictal tachycardia or bradycardia intensity | Through study completion, an average of 4 years
  Heart rate per minute
Abnormal heart-rate variability during the interictal period | Through study completion, an average of 4 years
  Inter bits per millisecond

CONTACTS AND LOCATIONS:
Locations (1):
- NeuroDigital@NeuroTech, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided